CLINICAL TRIAL: NCT05234671
Title: Exploring the Effects of a Combined Exercise Programme on Pain and Fatigue Outcomes in People With Systemic Sclerosis: A Large Multi-centre Randomised Controlled Trial
Brief Title: Exercise in People With Systemic Sclerosis
Acronym: SScPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Leiden University (Other); Rikshospitalet University Hospital (Other); Karolinska Institutet (Other); Aristotle University Of Thessaloniki (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ER35485474
Record Dates: First submitted 2022-01-14; First posted 2022-02-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The exercise group will perform a supervised combined (e.g., aerobic and resistance training) 12-week exercise programme, twice per week adjunct to the patient's standard care.
  Interventions: Other: Exercise programme
- Control group (No Intervention): The control group will not perform the exercise programme and will receive only the standard care.

INTERVENTIONS:
Other: Exercise programme — 12-week exercise programme. The estimated session's duration of 55 minutes. For the prescription of high intensity interval training (HIIT) and the collection of individualised peak power output (PPO) a baseline peak oxygen uptake on an arm crank ergometer will be performed. Each session will consist of 5 minutes warm up performing light to moderate intensity arm cranking (55-65% PPO), 30-minutes' high intensity interval training (HIIT; 30s 100% PPO/ 30s passive recovery) on an arm crank ergometer. The HIIT protocol will be combined with resistance training (RT) lasting for a total of 15 min.The intensity will be at 75-80% of one repetition maximum. Following each exercise session, patients will undertake a 5 min cool-down period.
  Arms: Exercise group

SUMMARY:
Raynaud's phenomenon and digital ulceration are two of the most common disease manifestations leading to digital and/or toe pain in systemic sclerosis (SSc). In addition to pain, fatigue has been identified as a key stressor and the most prevalent and debilitating symptom of SSc. Both, affect significantly quality of life (QoL) domains. Pharmacological therapeutic strategies have not been proved sufficiently effective in the management of SSc-induced pain and fatigue. Evidently the effectiveness of non-pharmacological interventions (e.g., exercise, cognitive behavioural therapy) is limited, although for some of them (i.e., exercise) evidence is promising. As yet, the effects of a feasible, long-term, tailored exercise programme on pain and fatigue in people with SSc have not been explored. Therefore, the investigators propose a multicentre (n=5) research clinical trial to assess the effect of a previously established, supervised 12-week combined (aerobic and resistance training) exercise programme on pain and fatigue. The 26-month study will recruit 180 people with SSc that will be allocated randomly to two groups. Group A will perform the exercise programme parallel to standard care and Group B will receive the standard care alone. All participants will be followed for 24-weeks. Results will inform clinical practice and may improve QoL for people with SSc.

DETAILED DESCRIPTION:
Background Pain in SSc originates from disease activity and is one of the most important patient-reported outcomes in rheumatology. It is estimated that up to 83% of people with SSc have significant pain. Raynaud's phenomenon (RP) and digital ulceration are two of the most common disease manifestations leading to digital and/or toe pain. Greater skin thickening is related to worse pain. SSc-related pain has been linked with numerous QoL domains, including mental health, physical health, and societal functioning (e.g., depression; with a strong relation between depression and pain, sleep, disability, fatigue, employment status. Given these personal, social, and financial implications for people with SSc, pain management should be one of the main goals of SSc-patient care. However, there is a lack of interventional research on SSc pain.

In addition to pain, fatigue has been identified as the main stressor and the most prevalent and debilitating symptom of SSc. Similar to pain, fatigue leads to a significant impairment of QoL, including physical disability, working, and parenting. In SSc, there is also a strong relation between fatigue and depression.

Pharmacological therapeutic strategies have been adopted in the management of pain and fatigue in SSc without being sufficiently effective. The evidence of the effectiveness of non-pharmacological interventions (e.g., the effects of exercise on SSc pain and fatigue) is limited, but promising. Engagement in regular exercise is associated with lower pain intensity and interference in people with SSc. Higher daily physical activity levels are associated with improved skin microvascular function in type 2 diabetes (a clinical condition with increased vasculopathy similar to that observed in SSc). This might explain partly why RP's pain is observed less in toes (as lower limbs are the most commonly used body part for daily activities) when compared to fingers. Thus, our focus would be mainly on digital pain in hands. Physically active people with SSc have lower levels of fatigue compared to inactive individuals. Moreover, evidence (e.g., one-to-one semi-structured interviews) from our recently completed feasibility study suggests that people with SSc feel more energetic and stronger following a combined (e.g., aerobic and resistance training) exercise programme, improving also their fitness and social life. Thus, a feasible, safe, long-term exercise programme for people with SSc that will improve pain and fatigue is warranted. Therefore, and being supported by published evidence, the investigators propose a multicentre RCT to assess the effect of such an exercise programme on pain and fatigue in this clinical population.

Research Objectives

* To investigate the effects of the proposed intervention on digital pain and fatigue of people with SSc.
* To investigate the effects of the proposed intervention on QoL, depression, cardiorespiratory fitness, strength of people with SSc.
* To investigate the effects of the proposed intervention on the digital structural vascular changes in people with SSc.

Research Plan/Methodology

Procedures Our RCT will recruit 180 people with SSc from five European study/recruitment centres (Sheffield Hallam University/Royal Hallamshire Hospital, UK; Karolinska Institutet/Sunderby Hospital, Sweden; Leiden University Medical Centre, Netherlands; Rigshospitalet, Copenhagen University, Copenhagen, Denmark; Aristotle University of Thessaloniki, Thessaloniki, Greece).

Experimental Design To further ensure high quality standards of the proposed intervention, the study's research manager will provide across centres standard operation procedure (SOP) digital manuals for all baseline measurements (including follow-up visits) and the delivery of the exercise programme, day-to-day quality monitoring, and an online video-meeting (consisting of two days) to demonstrate the delivery of a whole exercise session and all baseline measurements, and address any concerns of the co-investigators.

VISIT 1 (expected session duration: one hour; assessor blinded) Visit 1 baseline assessments will include anthropometrics, disease related clinical history (e.g., modified Rodnan skin score, Medsger disease severity score and digital ulcers history records). Pain, fatigue and QoL will be assessed via validated questionnaires. Structural changes in the microvascular lesions will be assessed via nailfold video-capillaroscopy. Peak power output (PPO; measured in watts) and cardiorespiratory fitness will be assessed via a peak oxygen uptake exercise test on an arm crank ergometer, and upper limb strength and endurance will be assessed via a hand grip and bicep curl tests. Patients will also complete a diary about their medical treatment history.

Randomisation- Management of Participants Following VISIT 1, participants will be randomised remotely (to ensure allocation and concealment) into Groups A (combined exercise) and B (control group), using a computer programme (nQuery Advisor 6.0, Statistical Solutions, Ireland) to generate stratified block-randomisation (by research centre, SSc-type, disease duration and severity), by an independent statistician.

Each participant will be allocated a unique trial number across all sites (e.g., SSc001) that will remain with them throughout the study. Patients will be free to withdraw at any point of the study without giving any reason and standard care for those patients will not be affected.

Intervention Following randomisation, Group A (combined exercise) will perform a 12-week exercise programme (aerobic and resistance training) twice per week. The exercise programme will be performed adjunct to standard care. Each session will consist of 5 minutes warm up performing light to moderate intensity arm cranking (55-65% PPO), 30-minutes' high intensity interval training (HIIT; 30s 100% PPO/ 30s passive recovery) on an arm crank ergometer. The HIIT protocol will be combined with resistance training (RT) lasting for a total of 15 min. RT will consist of an upper body circuit training (five exercises; Shoulder lateral raise in a sitting position, chest press on a bench in a 30° supine position; biceps curl and triceps extension in a sitting position, all exercises will be performed with dumbbells) for three circuits. The intensity will be at 75-80% of one repetition maximum (1-RM; that will be determined indirectly via validated 1-RM prediction formulas) performing 10 repetitions of each exercise interspersed by 20-30 s to allow for safe movement between exercises. The recovery period between circuits will last 2-3 min. Following each exercise session, patients will undertake a 5 min cool-down period, involving upper-limb light intensity aerobic exercise (e.g., corresponding to 'light intensity' based on rating of perceived exertion; RPE) and some light stretching. HR and RPE will be assessed at regular intervals throughout the supervised exercise session. Blood pressure (BP) will be assessed pre- and post-arm cranking and at the end of each session (duration: 45 minutes). Each session will be delivered as a one-to-one supervised session by a qualified health care professional (e.g., clinical exercise physiologist/physical therapist with experience in SSc) trainer. Group B will not perform the exercise programme and will receive the standard care. Following VISIT 3 (see below), Group B will be offered the same exercise intervention as in Group A. Any potential adverse events (e.g., pain) during the exercise sessions will be assessed for relation with the intervention and will be recorded by the health care professional. To support the successful participation of our participants, the investigators will use our "six pillars of adherence" framework (based upon "social support", "education", "reachability", "small groups intervention implementation", "reminders" and "simplicity"), which the investigators have used previously with excellent results in lifestyle interventions (i.e., over 90% of retention and 79% of completion).

VISITS 2, 3 (expected session duration: one hour; assessor-blinded) Three months (VISIT 2) and six months (VISIT 3) following VISIT 1, both Group A and Group B will repeat all the assessments. VISIT 2 will assess the effects of the exercise programme on study outcomes (e.g., pain and fatigue) immediately after the exercise intervention. VISIT 3 will examine whether any potential changes in pain and fatigue have been maintained in a long-term post-exercise intervention. Beside collecting data from the medical records, a detailed diary containing the medical prescriptions (drug name, dose, frequency) and any complications or disease exacerbations that might have occurred such as digital ulcers, hospitalisations (e.g., iloprost infusion) and / or amputations will be recorded by study researchers every three weeks via phone calls throughout the study for both groups.

Statistical analysis Data analysis will be performed as intention to treat, using SPSS software (IBM SPSS, New York, USA) and will be presented as mean ± SD. Normal distribution of the data and homogeneity of variances will be tested using the Shapiro-Wilk and Levene's test, respectively. The comparison between the two groups for pain and fatigue (primary outcomes) will be performed through independent t-tests and Chi-squared tests. Mixed model ANCOVA will also be performed to test the differences both within and between subject effects across time [three measurements: baseline, 12-week (primary time-point) and 24-week post baseline]. Effect sizes (Cohen's d) will be calculated wherever the results will be statistically significant with 0.2, 0.5, and 0.8 representing small, medium, and large effects respectively. Statistical significance will be set at p ≤ 0.05. Data analysis will commence at the end of the 2nd data collection post-baseline (i.e., 12-week).

Sample size calculation: the primary outcome was the RP pain. For the calculations a commercial software (G*Power 3.1.7, HHU of Düsseldorf) will be utilised by using data from two studies that examined the exercise training effects on SSc-QoL. Based on those calculations no more than 90 patients in each group (180 in total) will be needed to detect a difference in RP's pain at 3 months (significance level = 0.05; power =80%) accounting also for an estimated 15% dropout and 5% site effect.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Systemic Sclerosis according to the 2013 ACR/EULAR criteria experiencing Raynaud's phenomenon
* Age over 18 years old
* Ability to perform the prescribed exercise regime

Exclusion Criteria:

* Active disease-related exacerbations (e.g., active digital ulcers)
* Change of medical treatment (I.e., medical treatment which is related with the vascular function and blood flow such as calcium channel blockers and vasodilators) within the last 3 months (however, potential participants will be able to take part following that period)
* Advanced pulmonary involvement (e.g., pulmonary arterial hypertension)
* New York Heart Association class 3 or 4
* Inability to exercise
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Pain Assessment (Overall Pain) | 3-month follow up
  Overall pain will be assessed using the visual analogue scale (VAS) included in scleroderma health assessment questionnaire (SHAQ; VAS-SHAQ). VAS-SHAQ is consisted of a 15-cm which is converted to a continuous scale from 0 to 3 (1cm = 0.2 points on the VAS). For the VAS-SHAQ scale participants will be requested to self-complete the pain by placing a line perpendicular to the VAS line at the point that represents their overall and digital pain intensity.
Pain Assessment (Overall Pain) | 6-month follow up
  Overall pain will be assessed using the visual analogue scale (VAS) included in scleroderma health assessment questionnaire (SHAQ; VAS-SHAQ). VAS-SHAQ is consisted of a 15-cm which is converted to a continuous scale from 0 to 3 (1cm = 0.2 points on the VAS). For the VAS-SHAQ scale participants will be requested to self-complete the pain by placing a line perpendicular to the VAS line at the point that represents their overall and digital pain intensity.
Pain Assessment (Digital Pain) | 3-month follow up
  Digital pain will be assessed using a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases. The pain VAS will be comprised of a vertical line, usually 100 mm in length, anchored by 2 verbal descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst imaginable pain" (score of 100). For the digital VAS scale participants will be requested to self-complete the pain by placing a line perpendicular to the VAS line at the point that represents their overall and digital pain intensity.
Pain Assessment (Digital Pain) | 6-month follow up
  Digital pain will be assessed using a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases. The pain VAS will be comprised of a vertical line, usually 100 mm in length, anchored by 2 verbal descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst imaginable pain" (score of 100). For the digital VAS scale participants will be requested to self-complete the pain by placing a line perpendicular to the VAS line at the point that represents their overall and digital pain intensity.
Fatigue Assessment | 3-month follow up
  Fatigue in people with SSc will be assessed using the functional assessment of chronic illness therapy-fatigue (FACIT-F) which has also been utilised in studies assessing fatigue in people with SSc. Participants will be requested to self-complete this 40-item questionnaire which will assess fatigue and its impact on daily activities and function. FACIT-F is formatted in a Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much). All items contribute to the sum score with equal weight. The scale range is 0 to 52, with 0 being the worst possible score and 52 being the best possible score indicating no fatigue.
Fatigue Assessment | 6-month follow up
  Fatigue in people with SSc will be assessed using the functional assessment of chronic illness therapy-fatigue (FACIT-F) which has also been utilised in studies assessing fatigue in people with SSc. Participants will be requested to self-complete this 40-item questionnaire which will assess fatigue and its impact on daily activities and function. FACIT-F is formatted in a Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much). All items contribute to the sum score with equal weight. The scale range is 0 to 52, with 0 being the worst possible score and 52 being the best possible score indicating no fatigue.

SECONDARY OUTCOMES:
Quality of life questionnaire | 3-month follow up
  The systemic sclerosis quality of life (SScQoL) is a self-completed questionnaire comprising 29 questions exploring the impact of SSc on health and well-being, covering four themes identified by people with SSc: emotion, physical adaptation, impact on/with others and impact on self. It enables accurate evaluation of the impact of SSc on an individual or groups of people.
Quality of life questionnaire | 6-month follow up
  The systemic sclerosis quality of life (SScQoL) is a self-completed questionnaire comprising 29 questions exploring the impact of SSc on health and well-being, covering four themes identified by people with SSc: emotion, physical adaptation, impact on/with others and impact on self. It enables accurate evaluation of the impact of SSc on an individual or groups of people.
Depression scale questionnaire | 3-month follow up
  The Centre for Epidemiologic Studies-Depression Scale (CES-D) will be used to assess the depressive symptoms (which are associated with pain, fatigue and QoL). The CES-D has shown to be a reliable and valid measure of depressive symptoms in patients with SSc. The CES-D is a 20-item measure, with the frequency of each depressive symptom rated on a 4-point Likert scale ranging from 0 to 3 ("rarely or none of the time" to "most or all of the time").
Depression scale questionnaire | 6-month follow up
  The Centre for Epidemiologic Studies-Depression Scale (CES-D) will be used to assess the depressive symptoms (which are associated with pain, fatigue and QoL). The CES-D has shown to be a reliable and valid measure of depressive symptoms in patients with SSc. The CES-D is a 20-item measure, with the frequency of each depressive symptom rated on a 4-point Likert scale ranging from 0 to 3 ("rarely or none of the time" to "most or all of the time").
Microvascular assessment | 3-month follow up
  Nailfold video capillaroscopy (NVC) will be performed using an optical probe (100x and 200x contact lenses) connected to image analyse software. Images will be observed on a high-resolution colour monitor. Following 15 minutes of rest, NVC will be performed at a standardised room temperature of 20-22°C. The nailfolds of all 10 fingers will be examined in each patient, and a drop of immersion oil will be placed on the nailfold bed to improve the image resolution. Fingers that will be affected by severe local trauma will not be analysed. The following parameters will be recorded and analysed: presence of enlarged and giant capillaries, haemorrhages, loss of capillaries, disorganization of the vascular array, and ramified/bushy capillaries. A qualitative and semi-quantitative scoring of SSc patterns by NVC will be performed as described and validated previously
Microvascular assessment | 6-month follow up
  Nailfold video capillaroscopy (NVC) will be performed using an optical probe (200x contact lenses) connected to image analyse software. Images will be observed on a high-resolution colour monitor. Following 15 minutes of rest, NVC will be performed at a standardised room temperature of 20-25°C. The nailfolds of six digits (e.g., index, middle, and ring in both hands) will be examined in each patient, and a drop of immersion oil will be placed on the nailfold bed to improve the image resolution. Fingers that will be affected by severe local trauma will not be analysed. The following parameters will be recorded and analysed: presence of enlarged and giant capillaries, haemorrhages, loss of capillaries, disorganization of the vascular array, and ramified/bushy capillaries. A qualitative and semi-quantitative scoring of SSc patterns by NVC will be performed as described and validated previously
Peak oxygen uptake test on an arm crank ergometer | 3-month follow up
  Throughout the test gas exchange will be collected and analysed by an online breath-by-breath analysis system, and HR, BP and the electrocardiogram (ECG) will be continuously monitored. VO2peak will be defined as the average oxygen consumption during the final 30 s of exercise. The crank rate will be maintained above 50 rev min-1 (patient's will be allowed to select and maintain their own comfortable crank rate) and power requirements will be increased as a linear ramp at a rate of 10 W/min and 6 W/min for males and females, respectively. The test will be commenced with 3 min of warm-up (unloaded cranking). RPE ≥18 and/or inability to maintain a crank rate above 60 rev min-1 will be resulted in the termination of the test. After the exercise termination an unloaded bout of 2-3 min exercise at a crank rate below 50 rev min-1 will follow to allow for an active recovery period.
Peak oxygen uptake test on an arm crank ergometer | 6-month follow up
  Throughout the test gas exchange will be collected and analysed by an online breath-by-breath analysis system, and HR, BP and the electrocardiogram (ECG) will be continuously monitored. VO2peak will be defined as the average oxygen consumption during the final 30 s of exercise. The crank rate will be maintained above 50 rev min-1 (patient's will be allowed to select and maintain their own comfortable crank rate) and power requirements will be increased as a linear ramp at a rate of 10 W/min and 6 W/min for males and females, respectively. The test will be commenced with 3 min of warm-up (unloaded cranking). RPE ≥18 and/or inability to maintain a crank rate above 60 rev min-1 will be resulted in the termination of the test. After the exercise termination an unloaded bout of 2-3 min exercise at a crank rate below 50 rev min-1 will follow to allow for an active recovery period.
Handgrip strength test | 3-month follow up
  During the handgrip strength test the subject will hold the dynamometer on a seated position with the arm hanging by the side. The best of three attempts will be recorded.
Handgrip strength test | 6-month follow up
  During the handgrip strength test the subject will hold the dynamometer on a seated position with the arm hanging by the side. The best of three attempts will be recorded.
Biceps curl endurance test | 3-month follow up
  The biceps curl test will require the subject to repeatedly lift a 2kg weight (for women) or an 4kg weight (for men) for 30 seconds 60. The number of lifts will be recorded.
Biceps curl endurance test | 6-month follow up
  The biceps curl test will require the subject to repeatedly lift a 2kg weight (for women) or an 4kg weight (for men) for 30 seconds 60. The number of lifts will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Hallam University, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Ν/Α

REFERENCES:
- [Derived] Mitropoulos A, Jensen KY, Kouidi E, Bostrom C, Cuomo G, Diederichsen LP, Mattsson M, Hoekstra EM, De Vries-Bouwstra J, Dimitroulas T, Akil M, Jacobsen S, Klonizakis M; IMPACT-SSc CONSORTIUM. High-intensity interval and resistance training programme improves pain and fatigue outcomes in people with systemic sclerosis: a European multicentre randomised controlled trial. RMD Open. 2025 Nov 11;11(4):e005946. doi: 10.1136/rmdopen-2025-005946. PMID 41219127
- [Derived] Mitropoulos A, Bostrom C, Mattsson M, Kouidi E, Dimitroulas T, Liem SIE, Vlieland TPMV, de Vries-Bouwstra JK, Jacobsen S, Cuomo G, Akil M, Klonizakis M. Exploring the effects of a combined exercise programme on pain and fatigue outcomes in people with systemic sclerosis: study protocol for a large European multi-centre randomised controlled trial. Trials. 2022 Nov 28;23(1):962. doi: 10.1186/s13063-022-06853-1. PMID 36443836